CLINICAL TRIAL: NCT04043676
Title: Multicenter, Open-Label, Single Arm, Phase II Exploratory Study to Evaluate the Effect of a One-Year Consolidation Treatment With Ponatinib 15 mg on Treatment Free-Remission Rate in Patients With Philadelphia-Positive Chronic Myeloid Leukemia, Who Had Previously Achieved a Deep Molecular Response With Imatinib
Brief Title: Consolidation Treatment With Ponatinib 15 mg on Treatment Free-Remission Rate in Patients With Chronic Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Teófilo Hernando, Spain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PonaZero_study; 2017-004565-27 (EudraCT Number)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Leukemia; BCR-ABL positive; Myeloide; Philadelphia-positive; Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — ponatinib

STUDY DESIGN:
Intervention Model Description: 40 patients of both genders with chronic myeloid leukemia in MR4. Each patient will enter in the ponatinib consolidation phase (48 weeks) and them in the ponatinib treatment-free remission (96 weeks).
Masking Description: This is a single-arm, open label study designed to determine the rate of successful treatment free remission (TFR) in patients who achieved and maintained molecular response 4 (MR4) on ponatinib. This study has 2 main phases: ponatinib consolidation (48 weeks), and ponatinib TFR phases (96 weeks). All patients who have received a minimum of 4 years of imatinib therapy as unique TKI therapy, he/she has documented MR4 at least 12 months for study entry, and he/she shall continue with MR4 before the discontinuation of the ponatinib treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ponatinib Treatment (Experimental): Patients will be treated with 15 mg/day of ponatinib during 48 weeks. If a patient maintains MR4 throughout the 48 weeks, he/she will be eligible to start the ponatinib TFR phase. If a patient has confirmed loss of MR4 (two consecutive BCR-ABL > 0.01% IS) or loss of MMR (no confirmation needed), he/she will not be eligible for the TFR phase. Instead, he/she will restart imatinib treatment.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — All patient will take 15 mg/day ponatinib oral during 48 weeks.

SUMMARY:
Ponatinib has shown to induce deeper molecular responses compared with imatinib. Therefore, ponatinib treatment could increase the proportion of patients who could discontinue treatment successfully. This strategy that includes treatment change to a more powerful treatment before treatment discontinuation has not been evaluated in any of the previous clinical trials, and will be explored in the current study.

In this framework, the purpose is to determine the rate of successful treatment-free remission (TFR) within the first 48 weeks following cessation of treatment in patients who achieved Molecular Response 4 (MR4) on imatinib and maintained MR4 on ponatinib after a switch from imatinib. Eligible patients have been previously treated with imatinib as unique tyrosine kinase inhibitor (at least 4 years) and have documented MR4 (at least 12 months) at the time of switch to ponatinib to study entry.

DETAILED DESCRIPTION:
One decade ago, it was thought that cessation of Tyrosine Kinase Inhibitor (TKI) treatment in chronic myeloid leukemia in chronic phase (CML-CP) patients could be ineluctably followed by relapse, even in the setting of a complete molecular response. This paradigm was mainly based on two facts: the absence of the known graft vs leukemia effect of bone marrow transplant, and the demonstration that quiescent stem cells were resistant to TKI. Until then, the standard of care was to treat CML-CP patients indefinitely with TKI. The potential medical benefits of successful cessation include minimization of drug-drug interactions, elimination of chronic side effects, and pregnancy without exposure to TKIs. Hence, physicians, as well as patients, have shown a strong interest to explore cessation strategies for BCR-ABL inhibitors.

This paradigm of treating CML-CP patients with TKIs indefinitely was broken by the French "Stop imatinib study" (STIM), which investigated the feasibility of imatinib cessation in a highly selected group of patients who achieved and maintained complete molecular response (CMR) defined as undetectable BCR-ABL levels with high sample sensitivity (10-5 or greater) for a minimum of 2 years. With a median follow up of 30 months, 39% of patients have successfully stopped imatinib therapy. This provided the first evidence that achieving and maintaining deep molecular responses is a pre-requisite for successful therapy cessation.

Since the seminal study of the French Group, led by Mahon and Reiffers, multiple trials have studied the potential role of discontinuation of imatinib to achieve a stable TFR. Most of them required the absence of undetectable BCR-ABL to include the patient in the given study. In fact, the largest study of discontinuation, the EURO-SKI, and the ISAV study require a response MR4 or better to be eligible. Definition of relapse has also varied. In earlier studies, it was more stringent, and the trigger for reinitiating the treatment was the detection of the transcript. However, other studies have set the definition of relapse as the loss of major molecular response (MMR). The larger study in course, the EURO-SKI, has also defined the relapse as the loss of major molecular response. Taking all the studies together, the median probability of TFR by 2 years is 51%.

The experience is similar with patients treated with nilotinib upfront. The ENESTfreedom trial included 215 patients treated frontline with nilotinib having obtained a MR4.5, and receiving afterwards a consolidation phase with nilotinib 600 mg per day during one year. After this phase, those patients with stable MR4.5 discontinued the therapy. The results showed that the probability of TFR by 48 weeks was 51.6%.

Other trials have explored the possibility of a consolidation therapy with second-generation TKIs (2GTKI) in patients previously treated with imatinib. Some years ago, the ENESTcmr trial has shown that in patients not having achieved MR4.5, twice as many patients randomized to nilotinib vs. imatinib achieved MR4.5 after 12 months of treatment, allowing them to be eligible for discontinuation trials.

The rational of the ENESTop trial lies in this previous experience and explains its design: patients treated previously with imatinib, and having obtained a MR4.5 with nilotinib in second line, received a consolidation with nilotinib during 1 or 2 years, and then if the MR4.5 was stable, were eligible to discontinue therapy. With this strategy, the probability of TFR by 48 weeks was 58%. A similar approach has been followed by the Japanese investigators, but with patients having treated with dasatinib in second line. The probability of TFR by 2 years after discontinuation was 48%.

Response of Rescue Therapy after Relapse Patients after relapse were treated again, most of them with the TKI they received previous discontinuation. In the STIM study, in terms of regaining molecular response, 61 patients had a molecular recurrence, 56 regained undetectable BCR-ABL transcript level after a median of 4 months on imatinib (range 0-21 months). Five patients did not return to undetectable transcript level: four remained treatment-free with detectable transcript (range 0.05% to 0.3%) and one patient was switched to dasatinib due to loss of Complete Cytogenetic Response (CCyR). No loss of hematological response or progression to advanced phase was noted after stopping imatinib.

Similar results were observed in another study with a median 33 months of follow-up, and 55% of patients that met the protocol definition of molecular relapse (BCR-ABL detected by RT-qPCR in two consecutive tests). Twenty-one of 22 patients who restarted imatinib regained undetectable BCR-ABL transcript level. One patient remained in MMR at the 14-month follow-up.

Taking studies altogether the probability of regaining MMR is almost 100%, and the probability of regaining CMR ranges from 89%.

The rationale for the Study Design Ponatinib has shown to induce deeper molecular responses compared with imatinib. Therefore, ponatinib treatment could increase the proportion of patients who could discontinue treatment successfully. This strategy that includes treatment change to a more powerful treatment before treatment discontinuation has not been evaluated in any of the previous clinical trials, and will be explored in the current study.

In this framework, the purpose is to determine the rate of successful TFR within the first 48 weeks following cessation of treatment in patients who achieved MR4 on imatinib and maintained MR4 on ponatinib after a switch from imatinib. Eligible patients have been previously treated with imatinib as unique tyrosine kinase inhibitor (at least 4 years) and have documented MR4 (at least 12 months) at the time of switch to ponatinib to study entry.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. ECOG performance status of 0, 1, or 2.
3. Patient with diagnosis of BCR-ABL positive CML-CP.
4. Patient has received a minimum of 4 years of imatinib treatment, as unique TKI therapy.
5. Patient has achieved MR4 during at least 12 months with imatinib treatment, and determined by PCR lab assessment at screening.
6. Adequate end organ function.
7. Patients must have the following electrolyte values ≥ LLN limits or corrected to within normal limits with supplements prior to the first dose of study medication: Potassium, Magnesium, Total calcium (corrected for serum albumin).
8. Patients must have normal marrow function
9. Patients with preexisting, well-controlled, diabetes are not excluded.
10. Have normal QTcF interval on screening ECG evaluation, defined as QTcF of ≤ 450 ms in males or ≤ 470 ms in females.
11. Have a negative pregnancy test documented prior to enrollment
12. Be willing and able to comply with scheduled visits and study procedures.
13. Written informed consent obtained prior to any screening procedures.

Exclusion Criteria:

1. Prior AP, BC or autologous or allogenic transplant.
2. Patients with known atypical transcript.
3. CML treatment resistant mutation(s).
4. Are taking medications with a known risk of torsades de pointes (Appendix A)
5. Patient ever attempted to permanently discontinue imatinib or ponatinib treatment.
6. Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks.
7. Have clinically significant, uncontrolled, or active cardiovascular disease.
8. Have uncontrolled hypertension (diastolic blood pressure > 90 mmHg; systolic > 150 mmHg).
9. Have a history of alcohol abuse.
10. History of acute pancreatitis within 1 year prior to study entry or past medical history of chronic pancreatitis.
11. Have malabsorption syndrome or other gastrointestinal illness that could affect oral absorption of study drug.
12. Known presence of a significant congenital or acquired bleeding disorder unrelated to cancer.
13. Have a history of another malignancy; the exception is if patients have been disease-free for at least 5 years.
14. Have undergone surgery within 14 days prior to first dose of ponatinib.
15. Treatment with other investigational within 4 weeks of Day 1.
16. Patients actively receiving therapy with strong CYP3A4 inhibitors and/or inducers.
17. Patients actively receiving therapy with herbal medicines that are strong CYP3A4 inhibitors and/or inducers.
18. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval.
19. Have an ongoing or active infection.
20. Have a known history of human immunodeficiency virus infection.
21. Have hypersensitivity to the ponatinib active substance or to any of its inactive ingredients.
22. Pregnant or nursing (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Loss MR4 | 96 weeks (48 weeks ponatinib consolidation phase plus 48 weeks ponatinib treatment-free remission)
  Proportion of patients without confirmed loss of MR4 or loss of MMR (don't require confirmation) within 48 weeks following ponatinib therapy cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Luis Steegmann, MD PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Valentin Garcia Gutierrez, MD PhD, Principal Investigator — Hospital Universitario Ramon y Cajal; Rosa Ayala, MD PhD, Principal Investigator — Hospital Universitario Doce de Octubre; Luis Felipe Casado, Dr., Principal Investigator — Hospital Universitario Virgen del Rocio; Fermin Sanchez-Guijo, MD PhD, Principal Investigator — University of Salamanca; Juan Carlos Hernandez, Dr., Principal Investigator — Hospital Clínico Universitario de Valencia; Guillermo Orti, Dr., Principal Investigator — Hospital Vall d'Hebron; Blanca Xicoy, Dr., Principal Investigator — Hospital German Trials i Pujol; Antonio Jimenez, Dr., Principal Investigator — Hospital Regional Universitario de Malaga; Maria Teresa Gomez, Dr., Principal Investigator — Hospital Universitario de Gran Canarias Dr. Negrin
Locations (9):
- Spain (9):
  - Hospital Trials i Pujol, Badalona, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Universitario de Gran Canarias Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Unversitario de la Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Regional de Malaga, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Result] Graham SM, Jorgensen HG, Allan E, Pearson C, Alcorn MJ, Richmond L, Holyoake TL. Primitive, quiescent, Philadelphia-positive stem cells from patients with chronic myeloid leukemia are insensitive to STI571 in vitro. Blood. 2002 Jan 1;99(1):319-25. doi: 10.1182/blood.v99.1.319. PMID 11756187
- [Result] Hochhaus A, Masszi T, Giles FJ, Radich JP, Ross DM, Gomez Casares MT, Hellmann A, Stentoft J, Conneally E, Garcia-Gutierrez V, Gattermann N, Wiktor-Jedrzejczak W, le Coutre PD, Martino B, Saussele S, Menssen HD, Deng W, Krunic N, Bedoucha V, Saglio G. Treatment-free remission following frontline nilotinib in patients with chronic myeloid leukemia in chronic phase: results from the ENESTfreedom study. Leukemia. 2017 Jul;31(7):1525-1531. doi: 10.1038/leu.2017.63. Epub 2017 Feb 20. PMID 28218239
- [Result] Imagawa J, Tanaka H, Okada M, Nakamae H, Hino M, Murai K, Ishida Y, Kumagai T, Sato S, Ohashi K, Sakamaki H, Wakita H, Uoshima N, Nakagawa Y, Minami Y, Ogasawara M, Takeoka T, Akasaka H, Utsumi T, Uike N, Sato T, Ando S, Usuki K, Morita S, Sakamoto J, Kimura S; DADI Trial Group. Discontinuation of dasatinib in patients with chronic myeloid leukaemia who have maintained deep molecular response for longer than 1 year (DADI trial): a multicentre phase 2 trial. Lancet Haematol. 2015 Dec;2(12):e528-35. doi: 10.1016/S2352-3026(15)00196-9. Epub 2015 Nov 10. PMID 26686407
- [Result] Mahon FX, Rea D, Guilhot J, Guilhot F, Huguet F, Nicolini F, Legros L, Charbonnier A, Guerci A, Varet B, Etienne G, Reiffers J, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chroniques. Discontinuation of imatinib in patients with chronic myeloid leukaemia who have maintained complete molecular remission for at least 2 years: the prospective, multicentre Stop Imatinib (STIM) trial. Lancet Oncol. 2010 Nov;11(11):1029-35. doi: 10.1016/S1470-2045(10)70233-3. Epub 2010 Oct 19. PMID 20965785
- [Result] Mahon FX, Etienne G. Deep molecular response in chronic myeloid leukemia: the new goal of therapy? Clin Cancer Res. 2014 Jan 15;20(2):310-22. doi: 10.1158/1078-0432.CCR-13-1988. Epub 2013 Oct 28. PMID 24166905
- [Result] Mori S, Vagge E, le Coutre P, Abruzzese E, Martino B, Pungolino E, Elena C, Pierri I, Assouline S, D'Emilio A, Gozzini A, Giraldo P, Stagno F, Iurlo A, Luciani M, De Riso G, Redaelli S, Kim DW, Pirola A, Mezzatesta C, Petroccione A, Lodolo D'Oria A, Crivori P, Piazza R, Gambacorti-Passerini C. Age and dPCR can predict relapse in CML patients who discontinued imatinib: the ISAV study. Am J Hematol. 2015 Oct;90(10):910-4. doi: 10.1002/ajh.24120. Epub 2015 Sep 10. PMID 26178642
- [Result] Ross DM, Branford S, Seymour JF, Schwarer AP, Arthur C, Yeung DT, Dang P, Goyne JM, Slader C, Filshie RJ, Mills AK, Melo JV, White DL, Grigg AP, Hughes TP. Safety and efficacy of imatinib cessation for CML patients with stable undetectable minimal residual disease: results from the TWISTER study. Blood. 2013 Jul 25;122(4):515-22. doi: 10.1182/blood-2013-02-483750. Epub 2013 May 23. PMID 23704092
- [Result] Rousselot P, Charbonnier A, Cony-Makhoul P, Agape P, Nicolini FE, Varet B, Gardembas M, Etienne G, Rea D, Roy L, Escoffre-Barbe M, Guerci-Bresler A, Tulliez M, Prost S, Spentchian M, Cayuela JM, Reiffers J, Chomel JC, Turhan A, Guilhot J, Guilhot F, Mahon FX. Loss of major molecular response as a trigger for restarting tyrosine kinase inhibitor therapy in patients with chronic-phase chronic myelogenous leukemia who have stopped imatinib after durable undetectable disease. J Clin Oncol. 2014 Feb 10;32(5):424-30. doi: 10.1200/JCO.2012.48.5797. Epub 2013 Dec 9. PMID 24323036
- [Result] Lee SE, Choi SY, Bang JH, Kim SH, Jang EJ, Byeun JY, Park JE, Jeon HR, Oh YJ, Kim HJ, Kim YK, Park JS, Jeong SH, Kim SH, Zang DY, Oh S, Koo DH, Kim H, Do YR, Kwak JY, Kim JA, Kim DY, Mun YC, Mauro MJ, Kim DW. Predictive factors for successful imatinib cessation in chronic myeloid leukemia patients treated with imatinib. Am J Hematol. 2013 Jun;88(6):449-54. doi: 10.1002/ajh.23427. Epub 2013 Mar 28. PMID 23440689